CLINICAL TRIAL: NCT03299998
Title: Evaluation of Maxillary and Mandibulary Nerve Blocks on Morphine Consumption in Double-jaw Surgery, a Retrospective Study
Brief Title: Evaluation of Maxillary and Mandibulary Nerve Blocks on Morphine Consumption
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2017_001
Record Dates: First submitted 2017-09-14; First posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Dento Facial Dysmorphism
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BLOCK+: Patients who underwent maxillary and mandibulary block before surgery
  Interventions: Procedure: Maxillary and mandibular blocks; Procedure: General anesthesia
- BLOCK -: Patients who did not undergo maxillary and mandibulary block before surgery.
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: Maxillary and mandibular blocks — A Pajunk SonoPlex Stim needle 22G x 55 mm was used. For maxillary nerve block, needle was introduced next to the angle of the orbitae and the zygomatic ridge. The needle was sank until coming into contact of the temporal bone. It was then orientated to the controlateral nostril and sank of 1 cm. For mandibular block, needle was introduced in the pterygoid fossa under and perpendicularly to the zygomatic arch, and sank until the pterygoid process. The needle was then orientated towards controlateral orbitae and sank with neurostimulation. After a motor response at 0.6 milliampere (mA) and the disappearance of contraction at 0.3 mA, local mixture was injected. The mixing of local anesthesia was made of ropivacaine 5 mg/mL and clonidine 30 µg. Five mL were injected in every block for a total of 20 mL.
  Groups: BLOCK+
Procedure: General anesthesia — Anesthesia was standardized and provided using intravenous administration of propofol and remifentanil. Patients were mechanically ventilated with a mixture of air (50/50), and desflurane or sevoflurane, or Target-controlled infusion (TCI) propofol. One to 5 mg/kg of methyl-prednisolone were administered to reduce inflammatory response.

SUMMARY:
Background and Objectives: Double-jaw surgery is one of the most painful oral surgery, requiring multimodal analgesia including controlled morphine pump and its secondary effects. The aim of this study was to evaluate the effectiveness of face block (mandibulary and maxillary block analgesia) on the first 24 hours on morphine consumption in patients admitted for double jaw surgery.

DETAILED DESCRIPTION:
Methods: Patients undergoing double-jaw surgery between January 2015 and May 2017 were enrolled. Patients were separated into 2 groups: patients receiving maxillary-mandibulary nerve block and those no receiving it. The primary endpoint was the morphine consumption within 24 hours post-surgery. Secondary endpoints were the intra-operative remifentanil consumption, incidence of postoperative nausea and vomiting at 24 hours, morphine consumption in recovery room, length of stay in hospital.

ELIGIBILITY:
Inclusion Criteria:

- Male and female who underwent double jaw surgery

Exclusion Criteria:

* opposition to the study
* an additional surgical procedure
* preoperative consumption of morphine or derived from morphine
* perioperative N20

Age Groups: Child, Adult, Older Adult
Study Population: Male and female who underwent double jaw surgery
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
Cumulative morphine consumption within 24 hours post-surgery | 24 hours
  Cumulative morphine consumption measured using patient controlled analgesia (PCA-pump).

SECONDARY OUTCOMES:
Peroperative remifentanil consumption | End of surgery (2 hours in average)
  Remifentanil consumption in µg.kg-1 during surgery
Cumulative morphine consumption within 12 hours post-surgery | 12 hours
  Cumulative morphine consumption measured using patient controlled analgesia (PCA-pump).
Cumulative morphine consumption within 48 hours post-surgery | 48 hours
  Cumulative morphine consumption measured using patient controlled analgesia (PCA-pump).
Hospital length of stay | Up to hospital discharge (5 days in average)
  Delay between hospitalization date and date of hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No